CLINICAL TRIAL: NCT05868278
Title: The Effect of Interactive Learning Method on Nursing Students' Learning of Movement Needs: A Randomized Controlled Study
Brief Title: Interactive Learning Method in Nursing Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Yadigar Ordu, Principal Investigator, Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ErbakanU.
Record Dates: First submitted 2023-04-30; First posted 2023-05-22 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Learning, Spatial
MeSH Terms: conditions — Spatial Learning

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): It is the group in which the traditional learning method will be used.
- Experimental (Experimental): It is the group in which the interactive learning method will be used.
  Interventions: Other: Training method intervention

INTERVENTIONS:
Other: Training method intervention — Traditional learning method will be used in the control group. In the experimental group, interactive learning method will be used.
  Arms: Experimental

SUMMARY:
The research will be conducted to determine the effect of the interactive learning method on the learning of the movement requirement of nursing students. 192 first-year students enrolled in a nursing faculty in Turkey will form the universe. Students who meet the criteria for inclusion in the research will be randomly assigned to the experimental and control groups according to their academic achievement scores. It is envisaged that the research will be completed with approximately 160 students (80=experiment, 80=control). The data of the research will be collected with the "Descriptive Characteristics Form", "Movement Requirement Knowledge Test", "Case Analysis" and "Student Opinion Evaluation Form for Interactive Learning". Expert opinions are taken on the data collection forms. Necessary revisions will be made accordingly. A case for educational purposes This case example was prepared. This case study will be taught to the control group in the classroom with the traditional method. The same case study will be taught to the experimental group in the classroom with the interactive learning method. The Easytestmaker application will be used in the interactive learning method. The data collection forms will be applied to the groups in the form of pre-application and post-application. At the end of the research data will be analyzed.

DETAILED DESCRIPTION:
The introductory characteristics form consists of four closed-ended questions (age, gender, GPA, graduated high school) prepared to determine the demographic characteristics of the students. The movement requirement knowledge test consists of 15 questions, each of which has five options, prepared by the researchers in line with the literature in order to determine the students' knowledge levels about their movement needs. The questions were prepared in accordance with Bloom's taxonomy. In this context, considering that the students are in the first grade, three questions are for knowledge, three for comprehension, three for analysis, three for synthesis, and three for evaluation. After the test is prepared, it will be examined by a total of three experts, including a faculty member who is an expert in the field of Measurement and Evaluation and two faculty members who are experts in the field of Nursing Principles (1: Appropriate, 2: Appropriate but insufficient, 3: Not suitable). The concordance between expert opinions will be analyzed by Kendall's W test. Correct answers in the test will be evaluated as "10" points and wrong answers as "0" points. In this context, a minimum of "0" points and the highest "150" points can be obtained from the test. An increase in the score obtained from the test will show that the students' level of knowledge about movement needs is high. In the case analysis, correct answers given by the students will be evaluated as "10" points, and incorrect answers as "0" points. In this context, points will be made according to each correct and incorrect answer given by the students to the open-ended questions. An increase in the score will show that the students' case analysis skills for movement needs are high. The student opinion evaluation form on interactive learning was prepared by the researchers by scanning the literature in order to evaluate the opinions of the students in the experimental group about the interactive learning method. In this context, the form consists of 10 questions including five-point Likert-type scoring. After the theoretical training, the principal researcher will give the students an introductory feature form and will be asked to fill it in the classroom.Movement requirement knowledge test and evaluation case pre-test and post-test applications will be made. At the end of the study, students in the experimental group will be asked to fill in an evaluation form for the interactive learning method in order to get their opinions on the interactive learning method.

ELIGIBILITY:
Inclusion Criteria:

* Taking the Nursing Fundamentals course for the first time
* Volunteering to participate in research

Exclusion Criteria:

* Graduating from a health-related high school or university
* Difficulty speaking and understanding Turkish
* Not participating in theoretical training
* Not participating in group work
* Not participating in interactive learning
* Not filling out data collection forms wanting to leave research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-29 (Actual)

PRIMARY OUTCOMES:
The knowledge level of the students regarding the movement needs will be evaluated. | up to 1 month
  Evaluation will be in the form of a movement requirement knowledge test, an evaluation case, and a pre-test and post-test. Detailed information about data collection forms is given. After the post-test, the opinions of the students in the experimental group on interactive learning will be taken with the evaluation form.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Merkez, Konya, Turkey (Türkiye)

REFERENCES:
- [Derived] Ordu Y, Aydogan S, Caliskan N. The effect of interactive learning method on nursing students' learning of movement requirement: A randomized controlled study. Nurse Educ Today. 2024 Jun;137:106163. doi: 10.1016/j.nedt.2024.106163. Epub 2024 Mar 13. PMID 38503247